CLINICAL TRIAL: NCT02388906
Title: A Phase 3, Randomized, Double-blind Study of Adjuvant Immunotherapy With Nivolumab Versus Ipilimumab After Complete Resection of Stage IIIb/c or Stage IV Melanoma in Subjects Who Are at High Risk for Recurrence (CheckMate 238: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 238)
Brief Title: Efficacy Study of Nivolumab Compared to Ipilimumab in Prevention of Recurrence of Melanoma After Complete Resection of Stage IIIb/c or Stage IV Melanoma
Acronym: CheckMate 238
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-238; 2014-002351-26 (EudraCT Number)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ipilimumab and Placebo matching Nivolumab (Experimental)
  Interventions: Drug: Ipilimumab; Other: Placebo matching Nivolumab
- Nivolumab and Placebo matching Ipilimumab (Experimental)
  Interventions: Drug: Nivolumab; Other: Placebo matching Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Specified dose on specified days
  Arms: Ipilimumab and Placebo matching Nivolumab
Drug: Nivolumab — Specified dose on specified days
  Arms: Nivolumab and Placebo matching Ipilimumab
Other: Placebo matching Ipilimumab — Specified dose on specified days
  Arms: Nivolumab and Placebo matching Ipilimumab
Other: Placebo matching Nivolumab — Specified dose on specified days
  Arms: Ipilimumab and Placebo matching Nivolumab

SUMMARY:
The purpose of this study is to determine whether nivolumab is better than ipilimumab to prevent recurrence of melanoma.

ELIGIBILITY:
Inclusion Criteria:

* At least 15 years of age Except: where local regulations and/or institutional policies do not allow for subjects < 18 years of age (pediatric population) to participate. For those sites, the eligible subject population is ≥ 18 years of age
* Completely removed melanoma by surgery performed within 12 weeks of randomization
* Stage IIIb/C or Stage IV before complete resection
* No previous anti-cancer treatment

Exclusion Criteria:

* Ocular or uveal melanoma
* History of carcinomatosis meningitis
* History of auto-immune disease
* Treatment directed against the resected melanoma that is administrated after the surgery

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 906 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (136):
- United States (35):
  - Local Institution - 0036, Little Rock, Arkansas
  - Local Institution - 0117, La Jolla, California
  - Local Institution - 0189, Los Angeles, California
  - Local Institution - 0021, San Francisco, California
  - Local Institution - 0006, San Francisco, California
  - Local Institution - 0010, Aurora, Colorado
  - Local Institution - 0004, Washington D.C., District of Columbia
  - Local Institution - 0012, Jacksonville, Florida
  - Local Institution - 0019, Miami Beach, Florida
  - Local Institution - 0030, Orlando, Florida
  - Local Institution - 0032, Tampa, Florida
  - Local Institution - 0016, Atlanta, Georgia
  - Local Institution - 0106, Chicago, Illinois
  - Local Institution - 0013, Boston, Massachusetts
  - Local Institution - 0170, Boston, Massachusetts
  - Local Institution - 0171, Boston, Massachusetts
  - Local Institution - 0015, Ann Arbor, Michigan
  - Local Institution - 0002, Robbinsdale, Minnesota
  - Local Institution - 0017, St Louis, Missouri
  - Local Institution - 0123, Hackensack, New Jersey
  - Local Institution - 0095, New Brunswick, New Jersey
  - Local Institution - 0024, New York, New York
  - Local Institution - 0033, New York, New York
  - Local Institution - 0003, Charlotte, North Carolina
  - Local Institution - 0025, Durham, North Carolina
  - Local Institution - 0157, Columbus, Ohio
  - Local Institution - 0031, Portland, Oregon
  - Local Institution - 0029, Portland, Oregon
  - Local Institution - 0022, Allentown, Pennsylvania
  - Local Institution - 0001, Bethlehem, Pennsylvania
  - Local Institution - 0026, Charleston, South Carolina
  - Local Institution - 0014, Nashville, Tennessee
  - Local Institution - 0005, Dallas, Texas
  - Local Institution - 0027, Charlottesville, Virginia
  - Local Institution - 0126, Seattle, Washington
- Argentina (3):
  - Local Institution - 0142, Capital Federal, Buenos Aires
  - Local Institution - 0140, San Miguel de Tucumán, Tucumán Province
  - Local Institution, Córdoba
- Australia (10):
  - Local Institution - 0079, Gateshead, New South Wales
  - Local Institution - 0080, Westmead, New South Wales
  - Local Institution - 0078, Wollstonecraft, New South Wales
  - Local Institution - 0082, Greenslopes, Queensland
  - Local Institution - 0083, Southport, Queensland
  - Local Institution - 0084, Adelaide, South Australia
  - Local Institution - 0075, Heidelberg, Victoria
  - Local Institution - 0077, Prahran, Victoria
  - Local Institution - 0085, Nedlands, Western Australia
  - Local Institution - 0081, Camperdown
- Austria (2):
  - Local Institution - 0169, Graz
  - Local Institution - 0168, Salzburg
- Belgium (4):
  - Local Institution - 0038, Brussels
  - Local Institution - 0040, Brussels
  - Local Institution - 0037, Ghent
  - Local Institution - 0039, Leuven
- Canada (5):
  - Local Institution - 0051, Edmonton, Alberta
  - Local Institution - 0074, Vancouver, British Columbia
  - Local Institution - 0094, Toronto, Ontario
  - Local Institution - 0105, Montreal, Quebec
  - Local Institution - 0046, Québec, Quebec
- Czechia (4):
  - Local Institution - 0101, Hradec Králové
  - Local Institution - 0102, Ostrava-Poruba
  - Local Institution - 0099, Prague
  - Local Institution - 0100, Prague
- Finland (2):
  - Local Institution - 0047, Helsinki
  - Local Institution - 0048, Tampere
- France (6):
  - Local Institution - 0138, Lille
  - Local Institution - 0135, Marseille
  - Local Institution - 0134, Nantes
  - Local Institution - 0136, Paris
  - Local Institution - 0133, Pierre-Bénite
  - Local Institution - 0137, Toulouse
- Greece (2):
  - Local Institution - 0086, Athens
  - Local Institution - 0087, Neo Faliro
- Local Institution - 0163, Budapest, Hungary
- Ireland (4):
  - Local Institution - 0063, Dublin
  - Local Institution - 0166, Dublin
  - Local Institution - 0108, Dublin
  - Local Institution - 0064, Galway
- Italy (8):
  - Local Institution - 0112, Bergamo
  - Local Institution - 0116, Genova
  - Local Institution - 0115, Meldola (FC)
  - Local Institution - 0113, Milan
  - Local Institution - 0107, Napoli
  - Local Institution - 0111, Padua
  - Local Institution - 0114, Roma
  - Local Institution - 0110, Siena
- Japan (10):
  - Local Institution - 0179, Nagoya, Aichi-ken
  - Local Institution - 0161, Fukuoka, Fukuoka
  - Local Institution - 0174, Tsukuba, Ibaraki
  - Local Institution - 0162, Kumamoto, Kumamoto
  - Local Institution - 0160, Matsumoto, Nagano
  - Local Institution - 0175, Niigata, Niigata
  - Local Institution - 0176, Osaka, Osaka
  - Local Institution - 0159, Sunto-gun, Shizuoka
  - Local Institution - 0158, Chuo-ku, Tokyo
  - Local Institution - 0180, Chuo-shi, Yamanashi
- Netherlands (4):
  - Local Institution - 0042, Amsterdam
  - Local Institution - 0045, Groningen
  - Local Institution - 0043, Nijmegen
  - Local Institution - 0041, Veldhoven
- Norway (2):
  - Local Institution - 0098, Bergen
  - Local Institution - 0109, Oslo
- Poland (3):
  - Local Institution - 0150, Gdansk
  - Local Institution - 0149, Krakow
  - Local Institution - 0152, Warsaw
- Romania (2):
  - Local Institution - 0156, Craiova
  - Local Institution - 0153, Romania
- South Africa (5):
  - Local Institution - 0148, Johannesburg, Gauteng
  - Local Institution - 0145, Pretoria, Gauteng
  - Local Institution - 0147, Saxonwold, Johannesburg, Gauteng
  - Local Institution - 0181, Cape Town, Western Cape
  - Local Institution - 0146, Kraaifontein, Western Cape
- South Korea (4):
  - Local Institution - 0144, Songpa-gu, Seoul
  - Local Institution - 0129, Seoul
  - Local Institution - 0127, Seoul
  - Local Institution - 0128, Seoul
- Spain (4):
  - Local Institution - 0120, Barcelona
  - Local Institution - 0119, Madrid
  - Local Institution - 0121, Seville
  - Local Institution - 0122, Valencia
- Sweden (2):
  - Local Institution - 0050, Gothenberg
  - Local Institution - 0096, Lund
- Local Institution - 0167, Zurich, Switzerland
- Taiwan (3):
  - Local Institution - 0131, Kaohsiung City
  - Local Institution - 0132, Taichung
  - Local Institution - 0130, Taoyuan District
- United Kingdom (10):
  - Local Institution - 0057, Bristol, Avon
  - Local Institution - 0052, Swansea, Carmarthenshire
  - Local Institution - 0165, London, Greater London
  - Local Institution - 0054, Manchester, Greater Manchester
  - Local Institution - 0056, Southampton, Hampshire
  - Local Institution - 0177, Northwood, Middlesex
  - Local Institution - 0055, Oxford, Oxfordshire
  - Local Institution - 0060, Newcastle upon Tyne, Tyne and Wear
  - Local Institution - 0097, Leicester
  - Local Institution - 0053, Surrey

REFERENCES:
- [Derived] Ascierto PA, Del Vecchio M, Merelli B, Gogas H, Arance AM, Dalle S, Cowey CL, Schenker M, Gaudy-Marqueste C, Pigozzo J, Marquez-Rodas I, Butler MO, Di Giacomo AM, Gligich O, De La Cruz-Merino L, Arenberger P, Atkinson V, Nathan P, Hill A, Millward M, Fecher LA, Khushalani NI, Queirolo P, Soomro R, Rathod D, Askelson M, Pe Benito M, Joseph D, Larkin J. Nivolumab for Resected Stage III or IV Melanoma at 9 Years. N Engl J Med. 2025 Oct 18. doi: 10.1056/NEJMoa2504966. Online ahead of print. PMID 41124198
- [Derived] Weber JS, Middleton MR, Yates G, Sharpe DJ, Kurt M, Lobo M, Moshyk A, Vanderpuye-Orgle J, Mohr P. Estimating Long-Term Survivorship Rates Among Patients With Resected Stage III/IV Melanoma: Analyses From CheckMate 238 and European Organization for Research and Treatment of Cancer 18071 Trials. J Clin Oncol. 2025 Mar 10;43(8):929-937. doi: 10.1200/JCO.24.00237. Epub 2024 Oct 8. PMID 39378385
- [Derived] Weber J, Del Vecchio M, Mandala M, Gogas H, Arance AM, Dalle S, Cowey CL, Schenker M, Grob JJ, Chiarion-Sileni V, Marquez-Rodas I, Butler MO, Di Giacomo AM, de la Cruz-Merino L, Arenberger P, Atkinson V, Hill A, Fecher LA, Millward M, Khushalani NI, Queirolo P, Long GV, Lobo M, Askelson M, Ascierto PA, Larkin J. Outcomes With Postrecurrence Systemic Therapy Following Adjuvant Checkpoint Inhibitor Treatment for Resected Melanoma in CheckMate 238. J Clin Oncol. 2024 Nov;42(31):3702-3712. doi: 10.1200/JCO.23.01448. Epub 2024 Aug 5. PMID 39102624
- [Derived] Larkin J, Weber J, Del Vecchio M, Gogas H, Arance AM, Dalle S, Cowey CL, Schenker M, Grob JJ, Chiarion-Sileni V, Marquez-Rodas I, Butler MO, Di Giacomo AM, Middleton MR, De la Cruz-Merino L, Arenberger P, Atkinson V, Hill A, Fecher LA, Millward M, Khushalani NI, Queirolo P, Long GV, Lobo M, Askelson M, Ascierto PA, Mandala M. Adjuvant nivolumab versus ipilimumab (CheckMate 238 trial): Reassessment of 4-year efficacy outcomes in patients with stage III melanoma per AJCC-8 staging criteria. Eur J Cancer. 2022 Sep;173:285-296. doi: 10.1016/j.ejca.2022.06.041. Epub 2022 Aug 11. PMID 35964471
- [Derived] Weber JS, Ascierto PA, Middleton MR, Hennicken D, Zoffoli R, Pieters A, Amadi A, Kupas K, Kotapati S, Moshyk A, Schadendorf D. Indirect treatment comparison of nivolumab versus placebo as adjuvant treatment for resected melanoma. Eur J Cancer. 2021 Nov;158:225-233. doi: 10.1016/j.ejca.2021.08.028. Epub 2021 Oct 15. PMID 34663559
- [Derived] Mandala M, Larkin J, Ascierto PA, Del Vecchio M, Gogas H, Cowey CL, Arance A, Dalle S, Schenker M, Grob JJ, Chiarion-Sileni V, Marquez-Rodas I, Butler MO, Di Giacomo AM, Lutzky J, De La Cruz-Merino L, Atkinson V, Arenberger P, Hill A, Fecher L, Millward M, Khushalani NI, de Pril V, Lobo M, Weber J. Adjuvant nivolumab for stage III/IV melanoma: evaluation of safety outcomes and association with recurrence-free survival. J Immunother Cancer. 2021 Aug;9(8):e003188. doi: 10.1136/jitc-2021-003188. PMID 34452930
- [Derived] Ascierto PA, Del Vecchio M, Mandala M, Gogas H, Arance AM, Dalle S, Cowey CL, Schenker M, Grob JJ, Chiarion-Sileni V, Marquez-Rodas I, Butler MO, Maio M, Middleton MR, de la Cruz-Merino L, Arenberger P, Atkinson V, Hill A, Fecher LA, Millward M, Khushalani NI, Queirolo P, Lobo M, de Pril V, Loffredo J, Larkin J, Weber J. Adjuvant nivolumab versus ipilimumab in resected stage IIIB-C and stage IV melanoma (CheckMate 238): 4-year results from a multicentre, double-blind, randomised, controlled, phase 3 trial. Lancet Oncol. 2020 Nov;21(11):1465-1477. doi: 10.1016/S1470-2045(20)30494-0. Epub 2020 Sep 19. PMID 32961119
- [Derived] Weber J, Mandala M, Del Vecchio M, Gogas HJ, Arance AM, Cowey CL, Dalle S, Schenker M, Chiarion-Sileni V, Marquez-Rodas I, Grob JJ, Butler MO, Middleton MR, Maio M, Atkinson V, Queirolo P, Gonzalez R, Kudchadkar RR, Smylie M, Meyer N, Mortier L, Atkins MB, Long GV, Bhatia S, Lebbe C, Rutkowski P, Yokota K, Yamazaki N, Kim TM, de Pril V, Sabater J, Qureshi A, Larkin J, Ascierto PA; CheckMate 238 Collaborators. Adjuvant Nivolumab versus Ipilimumab in Resected Stage III or IV Melanoma. N Engl J Med. 2017 Nov 9;377(19):1824-1835. doi: 10.1056/NEJMoa1709030. Epub 2017 Sep 10. PMID 28891423
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 906 participants randomized and 905 treated. Reason for not treated: 1 participant withdrew consent.
Groups:
- Nivolumab 3 mg/kg: Nivolumab 3 mg/kg IV q2 wks and Ipilimumab placebo IV q3 wks for 4 doses then q12 wks starting at Wk 24
- Ipilimumab 10 mg/kg: Ipilimumab 10 mg/kg IV q3 wks for 4 doses then q12 wks starting at Wk 24 and Nivolumab placebo IV q2 wks
Period: Pre-Treatment Period
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Started (Started=Randomized) | 453 | 453
Completed (completed=treated) | 452 | 453
Not Completed | 1 | 0
Not completed — Participant withdrew consent | 1 | 0
Period: Treatment Period
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Started (Started=Treated) | 452 | 453
Completed (Completed=Finished the treatment period) | 275 | 123
Not Completed | 177 | 330
Not completed — Disease progression | 121 | 100
Not completed — Study drug toxicity | 41 | 208
Not completed — Adverse Event (AE) unrelated to study drug | 5 | 5
Not completed — Participant request to stop treatment | 5 | 9
Not completed — Participant withdrew consent | 2 | 3
Not completed — Poor/non-compliance | 0 | 1
Not completed — Participant no longer meets study criteria | 0 | 1
Not completed — Other reasons | 3 | 3

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg | Total
Number analyzed (Participants) | 453 | 453 | 906
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.34) | 53.6 (13.50) | 54.0 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 184 | 379
  Male | 258 | 269 | 527
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 215 | 208 | 423
  Unknown or Not Reported | 232 | 237 | 469
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 18 | 43
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 425 | 434 | 859
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS)
Description: RFS is defined as the time between the date of randomization and the date of first recurrence (local, regional or distant metastasis), new primary melanoma, or death (whatever the cause), whichever occurs first.
Time Frame: up to 36 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 453 | 453
Months | 52.37 [42.51 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 24.08 [16.56 to 35.09]
Statistical Analysis 1: Comparison: Nivolumab 3 mg/kg vs Ipilimumab 10 mg/kg; Test type: Superiority; p = 0.0003, Log Rank; Stratified log rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.60 to 0.86]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as as the time between the date of randomization and the date of death.
Time Frame: up to 106.6 months
Population: All randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 453 | 453
Months | NA [NA to NA] — Median not reached due to insufficient death events | NA [NA to NA] — Median not reached due to insufficient death events
Statistical Analysis 1: Comparison: Nivolumab 3 mg/kg vs Ipilimumab 10 mg/kg; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.88, 95.03% CI 2-sided [0.69 to 1.11] — Stratified Cox proportional hazard model

3. Secondary Outcome: The Safety and Tolerability of Nivolumab and Ipilimumab Measured by the Incidence of Adverse Events
Description: the safety and tolerability of Nivolumab and Ipilimumab was measured by the incidence of adverse events
Time Frame: reported between first dose and 30 days after last dose of study therapy
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 452 | 453
Participants
  Grade 3-4 | 116 | 251
  Any grade | 440 | 446

4. Secondary Outcome: The Safety and Tolerability of Nivolumab and Ipilimumab Measured by the Incidence of Serious Adverse Events
Description: The Safety and Tolerability of nivolumab and ipilimumab was measured by the incidence of serious adverse events
Time Frame: reported between the first dose and 30 days after last dose of study therapy
Population: all treated participants
Measure: Number; unit: Participants
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 452 | 453
Participants
  Grade 3-4 | 48 | 145
  Any grade | 80 | 184

5. Secondary Outcome: the Safety and Tolerability of Nivolumab and Ipilimumab Measured by the Incidence of Deaths
Description: the safety and tolerability of Nivolumab and Ipilimumab was measured by the incidence of Deaths
Time Frame: reported between first dose and 30 to 100 days after last dose of study therapy
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 452 | 453
Participants | 128 | 142

6. Secondary Outcome: The Safety and Tolerability of Nivolumab and Ipilimumab Measured by the Incidence of Laboratory Abnormalities
Description: The Safety and Tolerability of Nivolumab and Ipilimumab measured by the incidence of Laboratory abnormalities.
Time Frame: reported after first dose and within 30 days of last dose of the study therapy
Population: Participants with a CTC graded Laboratory Result for the given parameter from both Baseline and On-treatment
Measure: Number; unit: Participants
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 452 | 453
Participants
  Heamoglobin (grade1-4): number analyzed (Participants) | 447 | 440
  Heamoglobin (grade1-4) | 114 | 148
  Heamoglobin (Grade 3-4): number analyzed (Participants) | 447 | 440
  Heamoglobin (Grade 3-4) | 0 | 2
  Platelet count (grade1-4): number analyzed (Participants) | 447 | 440
  Platelet count (grade1-4) | 27 | 25
  Platelet count ( grade 3-4): number analyzed (Participants) | 447 | 440
  Platelet count ( grade 3-4) | 0 | 1
  Leukocytes (grade1-4): number analyzed (Participants) | 447 | 440
  Leukocytes (grade1-4) | 62 | 12
  Leukocytes (grade 3-4): number analyzed (Participants) | 447 | 440
  Leukocytes (grade 3-4) | 0 | 1
  Lymphocytes (grade1-4): number analyzed (Participants) | 446 | 439
  Lymphocytes (grade1-4) | 118 | 54
  Lymphocytes (grade 3-4): number analyzed (Participants) | 446 | 439
  Lymphocytes (grade 3-4) | 2 | 4
  Absolute Neutrophil count (Grade1-4): number analyzed (Participants) | 447 | 439
  Absolute Neutrophil count (Grade1-4) | 56 | 26
  Absolute Neutrophil count (Grade3-4): number analyzed (Participants) | 447 | 439
  Absolute Neutrophil count (Grade3-4) | 0 | 2
  Alkaline Phosphatase (grade1-4): number analyzed (Participants) | 441 | 437
  Alkaline Phosphatase (grade1-4) | 35 | 69
  Alkaline Phosphatase (Grade3-4): number analyzed (Participants) | 441 | 437
  Alkaline Phosphatase (Grade3-4) | 1 | 3
  Aspartate Aminotransferase (grade 1-4): number analyzed (Participants) | 445 | 440
  Aspartate Aminotransferase (grade 1-4) | 105 | 144
  Aspartate Aminotransferase(grade 3-4): number analyzed (Participants) | 445 | 440
  Aspartate Aminotransferase(grade 3-4) | 6 | 39
  Alkaline Aminotransferase (grade 1-4): number analyzed (Participants) | 447 | 443
  Alkaline Aminotransferase (grade 1-4) | 113 | 176
  Alkaline Aminotransferase(grade 3-4): number analyzed (Participants) | 447 | 443
  Alkaline Aminotransferase(grade 3-4) | 8 | 52
  Total Bilirubin (grade 1-4): number analyzed (Participants) | 446 | 439
  Total Bilirubin (grade 1-4) | 33 | 43
  Total Bilirubin (grade 3-4): number analyzed (Participants) | 446 | 439
  Total Bilirubin (grade 3-4) | 0 | 5
  Creatinine ( grade1-4): number analyzed (Participants) | 446 | 440
  Creatinine ( grade1-4) | 55 | 56
  Creatinine (grade 3-4): number analyzed (Participants) | 446 | 440
  Creatinine (grade 3-4) | 0 | 0
  Total Amylase ( grade1-4): number analyzed (Participants) | 400 | 392
  Total Amylase ( grade1-4) | 68 | 52
  Total Amylase (grade 3-4): number analyzed (Participants) | 400 | 392
  Total Amylase (grade 3-4) | 13 | 12
  Total Lipase ( grade1-4): number analyzed (Participants) | 438 | 427
  Total Lipase ( grade1-4) | 109 | 100
  Total Lipase (grade 3-4): number analyzed (Participants) | 438 | 427
  Total Lipase (grade 3-4) | 31 | 38
  Hypernatremia ( grade1-4): number analyzed (Participants) | 446 | 438
  Hypernatremia ( grade1-4) | 35 | 20
  Hypernatremia (grade 3-4): number analyzed (Participants) | 446 | 438
  Hypernatremia (grade 3-4) | 0 | 0
  Hyponatremia ( grade1-4): number analyzed (Participants) | 446 | 438
  Hyponatremia ( grade1-4) | 72 | 96
  Hyponatremia (grade 3-4): number analyzed (Participants) | 446 | 438
  Hyponatremia (grade 3-4) | 5 | 14
  Hyperkalemia ( grade1-4): number analyzed (Participants) | 445 | 439
  Hyperkalemia ( grade1-4) | 55 | 39
  Hyperkalemia (grade 3-4): number analyzed (Participants) | 445 | 439
  Hyperkalemia (grade 3-4) | 1 | 2
  Hypokalemia ( grade1-4): number analyzed (Participants) | 445 | 439
  Hypokalemia ( grade1-4) | 37 | 45
  Hypokalemia(grade 3-4): number analyzed (Participants) | 445 | 439
  Hypokalemia(grade 3-4) | 5 | 9
  Hypercalcemia ( grade1-4): number analyzed (Participants) | 434 | 422
  Hypercalcemia ( grade1-4) | 14 | 18
  Hypercalcemia(grade 3-4): number analyzed (Participants) | 434 | 422
  Hypercalcemia(grade 3-4) | 0 | 0
  Hypocalcemia ( grade1-4): number analyzed (Participants) | 434 | 422
  Hypocalcemia ( grade1-4) | 46 | 73
  Hypocalcemia(grade 3-4): number analyzed (Participants) | 434 | 422
  Hypocalcemia(grade 3-4) | 3 | 2
  Hypermagnesemia ( grade1-4): number analyzed (Participants) | 441 | 435
  Hypermagnesemia ( grade1-4) | 20 | 7
  Hypermagnesemia(grade 3-4): number analyzed (Participants) | 441 | 435
  Hypermagnesemia(grade 3-4) | 2 | 1
  Hypomagnesemia ( grade1-4): number analyzed (Participants) | 441 | 435
  Hypomagnesemia ( grade1-4) | 39 | 32
  Hypomagnesemia(grade 3-4): number analyzed (Participants) | 441 | 435
  Hypomagnesemia(grade 3-4) | 1 | 0

7. Secondary Outcome: Recurrence-free Survival by PD-L1 Expression
Description: Recurrence-free survival by PD-L1 Expression(5% tumor cell membrane expression)
Time Frame: up to 106.6 months
Population: All randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 453 | 453
Months
  Participants with >= 5% PD-L1 Expression,: number analyzed (Participants) | 153 | 154
  Participants with >= 5% PD-L1 Expression, | 70.41 [67.65 to 84.80] | 54.67 [24.15 to 84.40]
  Participants with < 5% PD-L1 Expression,: number analyzed (Participants) | 300 | 299
  Participants with < 5% PD-L1 Expression, | 38.677 [22.05 to 61.04] | 16.56 [11.14 to 26.51]
  Participants with Non-quantifiable PD-L1 Expression: number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Health Related Quality of Life (HRQoL) Evaluation
Description: HRQoL was measured by mean changes from baseline in EORTC-QLQ-C30 global health status/QoL composite scale and in remaining EORTC QLQ-C30 scales in all randomized participants.
  EORTC QLQ-C30 is the most commonly used QoL instrument in melanoma clinical studies, is a 30-item instrument that has gained wide acceptance in oncology clinical studies and comprises 5 functional scales (physical functioning, cognitive functioning, emotional functioning, social functioning and global quality of life) as well as nine symptom scales (fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Except for the overall health status and global quality of life items, responses for all items are 4 point categorical scales ranging from 1 (Not at all) to 4 (Very much). The overall health status/quality of life responses are 7-point Likert scales for which higher score reflects higher health status/quality of life for the 7-point Likert scale.
Time Frame: up to 36 months
Population: All randomized Participants with values from the second follow-up visit
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 334 | 308
Scores on a scale
  Physical functioning: number analyzed (Participants) | 327 | 307
  Physical functioning | -2.04 (15.134) | -4.88 (15.713)
  Role functioning: number analyzed (Participants) | 329 | 307
  Role functioning | -2.43 (25.219) | -3.85 (29.951)
  Emotional functioning: number analyzed (Participants) | 330 | 307
  Emotional functioning | 0.18 (20.282) | 1.43 (17.911)
  Cognitive functioning: number analyzed (Participants) | 330 | 307
  Cognitive functioning | -3.74 (18.364) | -4.67 (16.664)
  Social functioning: number analyzed (Participants) | 330 | 307
  Social functioning | -0.51 (22.085) | -3.53 (26.391)
  Global health status: number analyzed (Participants) | 330 | 307
  Global health status | -5.81 (20.046) | -7.00 (23.109)
  Fatigue: number analyzed (Participants) | 329 | 307
  Fatigue | 6.45 (21.605) | 9.05 (23.475)
  Nausea and vomiting: number analyzed (Participants) | 329 | 307
  Nausea and vomiting | 2.23 (12.622) | 1.90 (11.473)
  Pain: number analyzed (Participants) | 331 | 308
  Pain | 1.66 (23.314) | 4.38 (23.641)
  Dyspnea: number analyzed (Participants) | 328 | 306
  Dyspnea | 7.32 (22.741) | 5.45 (20.364)
  Insomnia: number analyzed (Participants) | 329 | 306
  Insomnia | 1.82 (28.692) | 3.05 (28.785)
  Appetite loss: number analyzed (Participants) | 328 | 307
  Appetite loss | 4.07 (22.660) | 2.61 (19.257)
  Constipation: number analyzed (Participants) | 329 | 307
  Constipation | 1.11 (17.904) | 0.33 (18.373)
  Diarrhea: number analyzed (Participants) | 330 | 306
  Diarrhea | 1.31 (20.831) | 3.38 (21.242)
  Financial difficulties: number analyzed (Participants) | 330 | 306
  Financial difficulties | -1.41 (23.348) | 0.54 (20.282)

9. Post Hoc Outcome: Recurrence-free Survival (RFS)
Description: as for outcome 1
Time Frame: up to 114 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 453 | 453
Months | 61.14 [42.87 to 89.23] | 24.15 [16.56 to 35.12]
Statistical Analysis 1: Comparison: Nivolumab 3 mg/kg vs Ipilimumab 10 mg/kg; Test type: Superiority; Log Rank; Stratified log rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.63 to 0.90]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): approximately up to 16 Months All-Cause mortality (From first dose to end of study): Approximately Up to 114 Months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Nivolumab 3 mg/kg | Ipilimumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 128/452 | 142/453
Serious Adverse Events (participants affected / at risk) | 106/452 | 215/453
Other Adverse Events (participants affected / at risk) | 421/452 | 438/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=452) | Ipilimumab 10 mg/kg (N=453)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 3
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 5
Adrenal suppression (Endocrine disorders) | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1
Hypophysitis (Endocrine disorders) | 3 | 18
Hypopituitarism (Endocrine disorders) | 0 | 1
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 5
Uveitis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Autoimmune colitis (Gastrointestinal disorders) | 0 | 5
Colitis (Gastrointestinal disorders) | 5 | 41
Diarrhoea (Gastrointestinal disorders) | 5 | 37
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 3
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Intussusception (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 2
Proctitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 0 | 1
Facial pain (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 8 | 11
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 2
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 7
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 3
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 2 | 0
Anorectal infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 7 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 3
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infected seroma (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 2
Meningitis aseptic (Infections and infestations) | 1 | 0
Mucormycosis (Infections and infestations) | 1 | 0
Myelitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 6
Pneumonia fungal (Infections and infestations) | 1 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Sinobronchitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 3
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Faecal volume increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
Liver function test increased (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Temporomandibular pain and dysfunction syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bell's palsy (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 4
Hypotonia (Nervous system disorders) | 0 | 1
IVth nerve disorder (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Miller Fisher syndrome (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Neurosarcoidosis (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Dependence (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 2
Giant cell arteritis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=452) | Ipilimumab 10 mg/kg (N=453)
Anaemia (Blood and lymphatic system disorders) | 13 | 26
Hyperthyroidism (Endocrine disorders) | 37 | 22
Hypophysitis (Endocrine disorders) | 6 | 42
Hypothyroidism (Endocrine disorders) | 53 | 35
Abdominal pain (Gastrointestinal disorders) | 53 | 78
Abdominal pain upper (Gastrointestinal disorders) | 33 | 21
Colitis (Gastrointestinal disorders) | 10 | 30
Constipation (Gastrointestinal disorders) | 47 | 46
Diarrhoea (Gastrointestinal disorders) | 171 | 250
Dry mouth (Gastrointestinal disorders) | 33 | 23
Dyspepsia (Gastrointestinal disorders) | 21 | 27
Nausea (Gastrointestinal disorders) | 110 | 135
Vomiting (Gastrointestinal disorders) | 39 | 68
Asthenia (General disorders) | 74 | 72
Chills (General disorders) | 11 | 31
Fatigue (General disorders) | 193 | 197
Influenza like illness (General disorders) | 32 | 39
Oedema peripheral (General disorders) | 24 | 29
Pyrexia (General disorders) | 39 | 105
Nasopharyngitis (Infections and infestations) | 53 | 24
Upper respiratory tract infection (Infections and infestations) | 43 | 32
Alanine aminotransferase increased (Investigations) | 38 | 88
Amylase increased (Investigations) | 29 | 26
Aspartate aminotransferase increased (Investigations) | 31 | 75
Blood alkaline phosphatase increased (Investigations) | 4 | 26
Lipase increased (Investigations) | 36 | 41
Weight decreased (Investigations) | 11 | 35
Decreased appetite (Metabolism and nutrition disorders) | 43 | 69
Arthralgia (Musculoskeletal and connective tissue disorders) | 103 | 80
Back pain (Musculoskeletal and connective tissue disorders) | 49 | 46
Myalgia (Musculoskeletal and connective tissue disorders) | 60 | 35
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 | 36
Dizziness (Nervous system disorders) | 47 | 39
Headache (Nervous system disorders) | 109 | 148
Anxiety (Psychiatric disorders) | 25 | 21
Insomnia (Psychiatric disorders) | 35 | 43
Cough (Respiratory, thoracic and mediastinal disorders) | 84 | 83
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 45
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 24 | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 | 37
Erythema (Skin and subcutaneous tissue disorders) | 31 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 136 | 179
Rash (Skin and subcutaneous tissue disorders) | 122 | 166
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27 | 52
Hypertension (Vascular disorders) | 33 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT02388906/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT02388906/SAP_001.pdf